CLINICAL TRIAL: NCT03104296
Title: Correlation Between Neonatal Cerebral Oxygenation and Later Psychomotor Outcome in Very-low-birth-weight Preterm Infants.
Brief Title: Correlation Between Cerebral Oxygenation and Neurodevelopment in VLBW Preterm Infants.
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2016-GQ; PRET_01_13 (Other: Ethic Committee of St. Orsola-Malpighi University Hospital); NIRS-SO (Other: Ethic Committee of St. Orsola-Malpighi University Hospital)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Psychomotor Impairment
Keywords: NIRS; Griffiths Mental Development Scales; prematurity
MeSH Terms: conditions — Psychomotor Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Griffiths Mental Development Scales — Griffiths Mental Development Scales investigate 5 main areas (locomotor, personal and social skills, hearing and language, eye and hand coordination, performance), providing a general developmental quotient (DQ) of infant's abilities and five sub-scale quotients (SQ) for each developmental area.
  The assessments are performed individually in a quiet room, over a 45-min period, by the same professional trained psychologist for the whole study period and are implemented in the presence of the infant's parent. The obtained results are adjusted for corrected age, in order to consider the neurobiological maturation of the enrolled infants.

SUMMARY:
The recent improvements in neonatal intensive care have led to a substantial increase in the survival rate of preterm infants; nevertheless, this population is still at high risk for long-term neurodevelopmental disabilities. Significant anatomical changes in brain structures and abnormal patterns of neuronal myelination and brain connectivity have been associated with preterm birth, with possible long-term effects on cognitive, motor and social skills.

The validation of clinical tools able to predict neurodevelopmental outcomes in the preterm population might help at identifying infants at greatest risk of impairment, who would benefit most from early supportive interventions exploiting brain neuroplasticity.

Near infrared reflected spectroscopy (NIRS) provides a bedside, non-invasive, continuous monitoring of cerebral oxygen saturation (CrSO2), which has been proposed as a predictive marker for later neurodevelopment in neonates undergone cardiac surgery; to date, however, evidence on the correlation between CrSO2 and later neurodevelopment in preterm infants is almost lacking.

This study aims to evaluate whether CrSO2 monitoring, performed before NICU discharge in clinically stable very low birth weight (VLBW) preterm infants, can predict psychomotor outcomes during the first 24 months of corrected age (ca).

DETAILED DESCRIPTION:
The improvements in neonatal intensive care occurred over the last decades have led to a substantial increase in the survival rate of preterm infants, especially of extremely low birth weight. Nevertheless, the delicate maturation of central nervous system (CNS) in the extrauterine environment, together with the possible development of prematurity-related clinical complications that could result in brain injury, place this population at high risk for long-term neurodevelopmental disabilities.

Significant anatomical changes in brain structures have been associated with preterm birth; among these, enlarged ventricles and subarachnoid spaces, reduced subcortical white matter and decreased cortical and deep nuclear grey matter are the most common. Additionally, there is increasing evidence of abnormal patterns of neuronal myelination and brain connectivity in preterm infants, with possible concerning long-term effects on language, motor and social skills. As for cognitive abilities, a direct correlation with gestational age (GA) has been previously shown in a large cohort of preterm born children at school age.

In its early phases, the developmental of CNS is characterized by an intrinsic neuroplasticity, according which repeated experiences could influence the arrangement of synaptic connections and neural circuitries, thus resulting in structural and functional changes. By exploiting this feature, an early establishment of supportive interventions¬ might aid to compensate the anatomical and functional constraints connected to preterm birth and to improve preterm infants' neurodevelopment.

The validation of clinical tools able to predict neurodevelopmental outcomes in the preterm population might help at identifying infants at greatest risk of impairment, who would benefit most from early rehabilitative interventions. Near infrared reflected spectroscopy (NIRS) provides a bedside, non-invasive, continuous monitoring of cerebral oxygen saturation (CrSO2) and has been largely adopted to assess neonatal brain oxygenation and perfusion in intensive care settings. Perioperative CrSO2 has been recently proposed as a possible predictor of later neurodevelopmental outcomes in neonates undergone cardiac surgery; data evaluating the correlation between CrSO2 and later neurodevelopment in preterm infants, however, are very scarce and limited to the first days of life; at this time, CrSO2 can be widely influenced by the occurrence of systemic haemodynamic instability and is blind to several clinical complications, known as potential causes of brain damage, that can occur later on during hospital stay and thus are not necessarily directly related to changes in cerebral oxygenation within the first days of life (e.g. necrotizing enterocolitis [NEC], late onset sepsis).

Hence, the aim of this study was to evaluate whether CrSO2 monitoring, performed before NICU discharge in clinically stable very low birth weight (VLBW) preterm infants, can predict psychomotor outcomes during the first 24 months of corrected age (ca).

Infants meeting eligibility criteria (for details see specific section) undergo a 3-hour continuous monitoring of CrSO2 by means of the INVOS 5100 oximeter when satisfying the following condition: stable clinical condition, no need for oxygen supplementation, full enteral feeding (defined as 160 ml/kg/day) After discharge, the enrolled infants are included in a long-term neurodevelopmental follow-up, which is part of the normal routine care for preterm-born infants and aims at the early identification and treatment of neurocognitive sequelae possibly related to preterm birth.

In this context, psychomotor outcome (PSO) is assessed at 6, 12, 18 and 24 months ca by means of the Griffiths Mental Development Scales 0-2 years [26]. These scales investigate five main areas (locomotor, personal and social skills, hearing and language, eye and hand coordination, performance), providing a general developmental quotient (DQ) of infant's abilities and five sub-scale quotients (SQ) for each of the developmental areas.

The Griffiths Scales are administered individually, over a 45-min period, by the same professional trained psychologist for the whole study period and are implemented in the presence of the infant's parent.

A correlation analysis between mean CrSO2 values and GQ/SQ scores at each follow-up appointment will be performed. In order to evaluate the effect of possible confounding variables on the observed results, a mixed model including a number of risk factors known to affect preterm infants' neurodevelopment will be built for hierarchical multiple regression analysis. Significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks
* birth weight <1500 g.

Exclusion Criteria:

* congenital abnormalities
* hypoxic-ischemic encephalopathy
* intraventricular haemorrhage grade 3-4
* post-haemorrhagic ventricular dilatation
* periventricular leukomalacia and/or porencephalic cysts
* general anaesthesia

Ages: 15 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to the Neonatal Intensive Care Unit (NICU) of St. Orsola-Malpighi Hospital, Bologna (Italy) fulfilling the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Psychomotor outcome | 24 months
  Psychomotor outcome is assessed by Griffiths Mental Development Scales 0-2 years. Psychomotor outcome is considered normal if DQ>88.6; lower values characterize psychomotor impairment, which is further defined as mild (-1 to -2 SD, corresponding to 88.6-76.9 DQ), moderate (-2 to -3 SD, corresponding to 76.8- 65.1 DQ) and severe (<-3 SD, corresponding to 65 DQ).

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Neonatologia, Day Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson DK, Chen J, Beare R, Adamson CL, Ellis R, Ahmadzai ZM, Kelly CE, Lee KJ, Zalesky A, Yang JYM, Hunt RW, Cheong JLY, Inder TE, Doyle LW, Seal ML, Anderson PJ. Structural connectivity relates to perinatal factors and functional impairment at 7years in children born very preterm. Neuroimage. 2016 Jul 1;134:328-337. doi: 10.1016/j.neuroimage.2016.03.070. Epub 2016 Apr 1. PMID 27046108
- [Background] Fischi-Gomez E, Vasung L, Meskaldji DE, Lazeyras F, Borradori-Tolsa C, Hagmann P, Barisnikov K, Thiran JP, Huppi PS. Structural Brain Connectivity in School-Age Preterm Infants Provides Evidence for Impaired Networks Relevant for Higher Order Cognitive Skills and Social Cognition. Cereb Cortex. 2015 Sep;25(9):2793-805. doi: 10.1093/cercor/bhu073. Epub 2014 May 2. PMID 24794920
- [Background] Sansavini A, Pentimonti J, Justice L, Guarini A, Savini S, Alessandroni R, Faldella G. Language, motor and cognitive development of extremely preterm children: modeling individual growth trajectories over the first three years of life. J Commun Disord. 2014 May-Jun;49:55-68. doi: 10.1016/j.jcomdis.2014.02.005. Epub 2014 Feb 22. PMID 24630591
- [Background] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166
- [Background] Sood ED, Benzaquen JS, Davies RR, Woodford E, Pizarro C. Predictive value of perioperative near-infrared spectroscopy for neurodevelopmental outcomes after cardiac surgery in infancy. J Thorac Cardiovasc Surg. 2013 Feb;145(2):438-445.e1; discussion 444-5. doi: 10.1016/j.jtcvs.2012.10.033. Epub 2012 Dec 6. PMID 23219333
- [Background] Verhagen EA, Van Braeckel KN, van der Veere CN, Groen H, Dijk PH, Hulzebos CV, Bos AF. Cerebral oxygenation is associated with neurodevelopmental outcome of preterm children at age 2 to 3 years. Dev Med Child Neurol. 2015 May;57(5):449-55. doi: 10.1111/dmcn.12622. Epub 2014 Nov 8. PMID 25382744